CLINICAL TRIAL: NCT03288493
Title: Open-Label, Multicenter, Phase 1 Study to Assess the Safety of P BCMA-101 in Subjects With Relapsed / Refractory Multiple Myeloma (MM) Followed by a Phase 2 Assessment of Response and Safety (PRIME)
Brief Title: P-BCMA-101 Tscm CAR-T Cells in the Treatment of Patients With Multiple Myeloma (MM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase I portion of the study was completed. The phase II portion of the study was terminated early to focus on an Allogeneic BCMA CAR-T program.
Sponsor: Poseida Therapeutics, Inc. (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P-BCMA-101-001
Record Dates: First submitted 2017-09-13; First posted 2017-09-20 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: CAR-T cells
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Phase 1: open label, 3 + 3 design of dose-escalating cohorts Phase 2: open label, administered as a total dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 1: P-BCMA-101 CAR-T cells (Experimental): Single ascending dose cohorts, given in a single intravenous infusion of CAR-T cells. Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-101 CAR-T cells; Drug: Rimiducid
- Phase 1 P-BCMA-101 CAR-T cells (Cohort A) (Experimental): Single dose given across two intravenous infusions of CAR-T cells. Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-101 CAR-T cells; Drug: Rimiducid
- Phase 1 P-BCMA-101 CAR-T cells (Cohort B) (Experimental): Single dose given across three intravenous infusions of CAR-T cells. Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-101 CAR-T cells; Drug: Rimiducid
- Phase 1 P-BCMA-101 CAR-T cells (Cohort C) (Experimental): Single dose given across two intravenous infusions of CAR-T cells. Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-101 CAR-T cells; Drug: Rimiducid
- Phase 1 P-BCMA-101 CAR-T cells with Comb.Therapy (Cohort R) (Experimental): Single intravenous infusion of CAR-T cells, with combination therapy, beginning one week before CAR-T infusion. Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-101 CAR-T cells; Drug: Rimiducid
- Phase 1 P-BCMA-101 CAR-T cells with Comb.Therapy (Cohort RP) (Experimental): Single intravenous infusion of CAR-T cells, with combination therapy, beginning one week before apheresis. Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-101 CAR-T cells; Drug: Rimiducid
- Phase 1 P-BCMA-101 CAR-T cells with Comb.Therapy (Cohort RIT) (Experimental): Single intravenous infusion of CAR-T cells, with combination therapy, beginning one week before CAR-T infusion. Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-101 CAR-T cells; Drug: Rimiducid
- Phase 2: P-BCMA-101 CAR-T Cells (Experimental): CAR-T cells administered via intravenous infusion as a total dose
  Interventions: Biological: P-BCMA-101 CAR-T cells; Drug: Rimiducid

INTERVENTIONS:
Biological: P-BCMA-101 CAR-T cells — P-BCMA-101 is an autologous, principally Tscm, CAR-T cell product (also called called a CARTyrin T cell product) targeting the myeloma selective protein BCMA. P-BCMA-101 cells are produced using a non-viral vector carrying the gene for an anti-BCMA Centyrin-based (small, fully human binding domain, designed to increase T cell persistence and decrease exhaustion) chimeric antigen receptor (CAR). Secondary to the large carrying capacity of the non-viral vector, P-BCMA-101 cells carry two additional genes, a selection gene used to manufacture a purified product and a "safety switch" gene to allow the cells to be eliminated if desired. Rimiducid (safety switch activator) may be administered as indicated.
Drug: Rimiducid — Rimiducid (safety switch activator) may be administered as indicated.

SUMMARY:
Phase 1 of the study is comprised of an open-label, single ascending dose (SAD), multiple cohort study; a multiple dose cycle administration cohort study; and a combination administration study of P-BCMA-101 autologous T stem cell memory (Tscm) CAR-T cells in patients with relapsed / refractory MM. Followed by a Phase 2, open-label, efficacy and safety study. Rimiducid may be administered as indicated.

DETAILED DESCRIPTION:
Phase 1 follows a 3 + 3 design of dose-escalating cohorts. Phase 2 of the study is an open-label multi-center efficacy and safety study. After a patient enrolls, leukapheresis will be performed to obtain peripheral blood mononuclear cells which will be sent to a manufacturing site to produce P-BCMA-101 CAR-T cells. The cells will then be returned to the investigational site and, after a standard chemotherapy based conditioning regimen, will be administered to the patient across 1-3 infusions, with or without combination therapy. Treated patients will undergo serial measurements of safety, tolerability and response. Rimiducid may be administered as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ≥18 years of age
* Must have a confirmed diagnosis of active MM
* Must have measurable MM
* Must have relapsed / refractory MM, having received treatment with proteasome inhibitor and IMiD [Phase 2: Must have relapsed / refractory MM, and refractory to last line of therapy, having received treatment with proteasome inhibitor, an IMiD, CD38 targeted therapy and undergone autologous stem cell transplant (ASCT) or not a candidate for ASCT.]
* Must have adequate hepatic, renal, cardiac and hematopoietic function

Exclusion Criteria:

* Is pregnant or lactating
* Has inadequate venous access and/or contraindications to leukapheresis
* Has active hemolytic anemia, plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome, disseminated intravascular coagulation, leukostasis, amyloidosis, significant autoimmune, CNS or other malignant disease
* Has an active second malignancy (not disease-free for at least 5 years) in addition to MM, excluding low-risk neoplasms such as non-metastatic basal cell or squamous cell skin carcinoma.
* Has active autoimmune disease
* Has a history of significant central nervous system (CNS) disease, such as stroke, epilepsy, etc.
* Has an active systemic infection
* Has hepatitis B or C virus, human immunodeficiency virus (HIV), or human T-lymphotropic virus (HTLV) infection, or any immunodeficiency syndrome.
* Has any psychiatric or medical disorder that would preclude safe participation in and/or adherence to the protocol
* Has receiving immunosuppressive or other contraindicated therapies within the excluded time frame from entry
* Has CNS metastases or symptomatic CNS involvement
* Has a history of having undergone allogeneic stem cell transplantation, or any other allogeneic or xenogeneic transplant, or has undergone autologous transplantation within 90 days.
* Unable to take acetylsalicylic acid (ASA) daily as prophylactic anticoagulation. (Cohorts R and RP only).
* History of thromboembolic disease within the past 6 months, regardless of anticoagulation (Cohorts R and RP only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Belani, M.D., Study Director — Sponsor Executive Medical Director
Locations (16):
- United States (16):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of California Davis, Davis, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Wayne State - Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center, Hackensack, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington

REFERENCES:
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: P-BCMA-101 CAR-T Cells: Single administration dose cohorts, given in a single intravenous infusion of CAR-T cells. Rimiducid may be administered as indicated.
- Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort R): Single intravenous infusion of CAR-T cells, with combination therapy, beginning one week before CAR-T infusion.
Period: Overall Study
Arm/Group | Phase 1: P-BCMA-101 CAR-T Cells | Phase 1 P-BCMA-101 CAR-T Cells (Cohort A) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort B) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort R) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RP) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RIT) | Phase 2: P-BCMA-101 CAR-T Cells
Started | 69 | 3 | 1 | 8 | 5 | 16 | 3
Completed (Completed Study is defined as a subject completing Post-Treatment Follow-up Visits to Month 24.) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 66 | 3 | 1 | 8 | 5 | 16 | 3
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Significant progression of malignancy requiring alternative, medical, radiation or surgical interven | 52 | 3 | 1 | 6 | 5 | 10 | 3
Not completed — Termination of the study by the PI, the sponsor, the study funder, the IRB/IEC or the FDA | 6 | 0 | 0 | 2 | 0 | 4 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — other reason not listed above | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: P-BCMA-101 CAR-T Cells | Phase 1 P-BCMA-101 CAR-T Cells (Cohort A) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort B) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort R) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RP) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RIT) | Phase 2: P-BCMA-101 CAR-T Cells | Total
Number analyzed (Participants) | 69 | 3 | 1 | 8 | 5 | 16 | 3 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 2 | 1 | 5 | 3 | 8 | 2 | 60
  >=65 years | 30 | 1 | 0 | 3 | 2 | 8 | 1 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 0 | 1 | 4 | 2 | 7 | 2 | 39
  Male | 46 | 3 | 0 | 4 | 3 | 9 | 1 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 0 | 0 | 1 | 1 | 0 | 7
  Not Hispanic or Latino | 60 | 3 | 1 | 8 | 3 | 14 | 3 | 92
  Unknown or Not Reported | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 1 | 0 | 2 | 0 | 3 | 1 | 20
  White | 48 | 1 | 1 | 6 | 3 | 10 | 2 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 0 | 0 | 0 | 2 | 2 | 0 | 11
Region of Enrollment [Number; unit: participants]
  United States | 69 | 3 | 1 | 8 | 5 | 16 | 3 | 105

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Assess the Safety of P-BCMA-101
Description: Incidence and severity of treatment-emergent adverse events
Time Frame: Baseline through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: P-BCMA-101 CAR-T Cells | Phase 1 P-BCMA-101 CAR-T Cells (Cohort A) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort B) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort R) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RP) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RIT)
Number analyzed (Participants) | 67 | 3 | 1 | 8 | 5 | 16
Participants
  TEAE Related to P-BCMA-101 | 56 | 3 | 0 | 7 | 2 | 13
  TEAE Not Related to P-BCMA-101 | 11 | 0 | 1 | 1 | 3 | 3

2. Primary Outcome: Phase 1: Maximum Tolerated Dose of P-BCMA-101
Description: Rate of dose limiting toxicities (DLT)
Time Frame: Baseline through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: P-BCMA-101 CAR-T Cells | Phase 1 P-BCMA-101 CAR-T Cells (Cohort A) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort B) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort R) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RP) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RIT) | Phase 2: P-BCMA-101 CAR-T Cells
Number analyzed (Participants) | 69 | 3 | 1 | 8 | 5 | 16 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | NA — DLT not applicable for Phase 2 participants

3. Primary Outcome: Phase 2: Assess the Safety of P-BCMA-101
Description: Incidence and severity of treatment-emergent adverse events
Time Frame: Baseline through 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: P-BCMA-101 CAR-T Cells
Number analyzed (Participants) | 3
Participants
  TEAE Related to P-BCMA-101 | 2
  TEAE Not Related to P-BCMA-101 | 1

4. Primary Outcome: Phase 2: Assess the Efficacy of P-BCMA-101 (ORR)
Description: According to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma:
  Overall Response Rate (ORR)-Percentage of patients with complete response (CR), very good partial response (VGPR), or partial response (PR).
Time Frame: Baseline through 24 months
Population: Independent Review Committee (IRC) was not formed to assess ORR as the Phase II portion of the study was terminated early to focus on an Allogeneic BCMA CAR-T program.
Arm/Group | Phase 2: P-BCMA-101 CAR-T Cells
Number analyzed (Participants) | 0

5. Primary Outcome: Phase 2: Assess the Efficacy of P-BCMA-101 (DOR)
Description: According to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma:
  Duration of Response (DOR)-Time from complete response (CR), very good partial response (VGPR), or partial response (PR) to progressive disease.
Time Frame: Baseline through 24 months
Population: Independent Review Committee (IRC) was not formed to assess DOR as the Phase II portion of the study was terminated early to focus on an Allogeneic BCMA CAR-T program.
Arm/Group | Phase 2: P-BCMA-101 CAR-T Cells
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 1:Assess the Safety of P-BCMA-101
Description: Incidence and severity of treatment-emergent adverse events
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

7. Secondary Outcome: Phase 1:Assess the Feasibility P-BCMA-101
Description: Ability to generate protocol-prescribed doses of P-BCMA-101.
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

8. Secondary Outcome: Phase 1: Anti-myeloma Effect of P-BCMA-101 (ORR)
Description: as for outcome 4
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

9. Secondary Outcome: Phase 1: Anti-myeloma Effect of P-BCMA-101 (TTR)
Description: According to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma:
  Time to Response (TTR)-Time to complete response (CR), very good partial response (VGPR), or partial response (PR) to progressive disease.
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

10. Secondary Outcome: Phase 1: Anti-myeloma Effect of P-BCMA-101 (DOR)
Description: as for outcome 5
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

11. Secondary Outcome: Phase 1: Anti-myeloma Effect of P-BCMA-101 (PFS)
Description: According to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma:
  Progression Free Survival (PFS)-Time from P-BCMA-101 treatment to progressive disease.
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

12. Secondary Outcome: Phase 1: Anti-myeloma Effect of P-BCMA-101 (OS)
Description: According to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma:
  Overall Survival (OS)-Duration of survival from time of treatment with P-BCMA-101.
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

13. Secondary Outcome: Phase 1: The Effect of Cell Dose to Guide Selection of Doses for Further Assessment in Phase 2/3 Studies
Description: Incidence and severity of CRS events graded using Lee criteria (Lee, 2014)
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

14. Secondary Outcome: Phase 2: Incidence and Severity of Cytokine Release Syndrome (CRS)
Description: Incidence and severity of CRS events graded using Lee criteria (Lee, 2014)
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

15. Secondary Outcome: Phase 2: Evaluate Efficacy Endpoints (IL-6)
Description: Rate of IL-6 antagonist
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

16. Secondary Outcome: Phase 2: Evaluate Efficacy Endpoints (C)
Description: Corticosteroid Use
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

17. Secondary Outcome: Phase 2: Evaluate Efficacy Endpoints (R)
Description: Rimiducid Use
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

18. Secondary Outcome: Phase 2: Evaluate Efficacy Endpoints (OS)
Description: as for outcome 12
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

19. Secondary Outcome: Phase 2: Evaluate Efficacy Endpoints (PFS)
Description: as for outcome 11
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

20. Secondary Outcome: Phase 2: Evaluate Efficacy Endpoints (TTR)
Description: as for outcome 9
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

21. Secondary Outcome: Phase 2: Evaluate Efficacy Endpoints (MRD)
Description: Minimum residual disease negative rate
Time Frame: Baseline through Month 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through Month 24
Description: Treatment-emergent adverse events (TEAEs) are protocol-defined AEs that occur from the date of P-BCMA-101 infusion until study completion or subject withdrawal from study. Coded to system organ class and preferred term.
Groups:
- Retreatment: If a subject's disease progressed and sufficient P-BCMA-101 cells were available from initial manufacturing, a subject may have received an additional P-BCMA-101 infusion at up to the highest dose level that had completed DLT assessment.
Arm/Group | Phase 1: P-BCMA-101 CAR-T Cells | Phase 1 P-BCMA-101 CAR-T Cells (Cohort A) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort B) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort R) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RP) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RIT) | Phase 2: P-BCMA-101 CAR-T Cells | Retreatment
All-Cause Mortality (participants affected / at risk) | 23/69 | 0/3 | 0/1 | 3/8 | 1/5 | 0/16 | 1/3 | 2/5
Serious Adverse Events (participants affected / at risk) | 39/69 | 1/3 | 1/1 | 7/8 | 2/5 | 6/16 | 2/3 | 2/5
Other Adverse Events (participants affected / at risk) | 63/69 | 3/3 | 1/1 | 7/8 | 5/5 | 16/16 | 3/3 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: P-BCMA-101 CAR-T Cells (N=69) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort A) (N=3) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort B) (N=1) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort R) (N=8) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RP) (N=5) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RIT) (N=16) | Phase 2: P-BCMA-101 CAR-T Cells (N=3) | Retreatment (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (17) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia adenoviral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 6 (6) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: P-BCMA-101 CAR-T Cells (N=69) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort A) (N=3) | Phase 1 P-BCMA-101 CAR-T Cells (Cohort B) (N=1) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort R) (N=8) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RP) (N=5) | Phase 1 P-BCMA-101 CAR-T Cells With Comb.Therapy (Cohort RIT) (N=16) | Phase 2: P-BCMA-101 CAR-T Cells (N=3) | Retreatment (N=5)
Neutropenia (Blood and lymphatic system disorders) | 48 (189) | 3 (8) | 0 (0) | 3 (6) | 5 (12) | 13 (32) | 2 (2) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 32 (132) | 3 (4) | 0 (0) | 5 (8) | 2 (3) | 6 (8) | 2 (4) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 33 (92) | 1 (1) | 1 (1) | 2 (5) | 3 (5) | 5 (10) | 2 (2) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 20 (49) | 3 (6) | 1 (1) | 3 (5) | 1 (1) | 6 (10) | 2 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 25 (33) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 19 (23) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 6 (7) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 14 (18) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (12) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 22 (27) | 2 (2) | 0 (0) | 5 (7) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 19 (26) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 8 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 18 (22) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (30) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 15 (29) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 11 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (8) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (10) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (15) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT03288493/Prot_SAP_000.pdf